CLINICAL TRIAL: NCT03879265
Title: Validation of a Noninvasive Chromosome Screening (NICS) Method Using the Culture Medium
Brief Title: Validation of a NICS Method Using the Culture Medium
Status: Completed | Type: Observational
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Belen Lledo, Principal investigator, Instituto Bernabeu
Other Study IDs: IBB11
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Chromosome Abnormality; Abnormality
Keywords: Diagnosis; Reproduction; Chromosomal Endowment
MeSH Terms: conditions — Chromosome Aberrations; Congenital Abnormalities; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Embryo culture medium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: No intervention. Couples who come to the study center to carry out a PGT-A cycle will be selected. Only couples that will use their own gametes will be selected and the indication of PGT-A will be advanced maternal age, failure of implantation, repeat abortion, male factor or structural chromosomal alterations. The results of chromosomal status of the embryo will be compared using the NICS and the conventional invasive method (PGT-A).
  Interventions: Diagnostic Test: Noninvasive chromosome screening

INTERVENTIONS:
Diagnostic Test: Noninvasive chromosome screening — Screening based on MALBAC-NGS technology

SUMMARY:
This study aims to validate a non-invasive method of chromosomal screening (NICS), based on the Multiple Annealing and Looping Based Amplification Cycles- Next-generation Sequencing (MALBAC-NGS) technology, in order to determine the chromosomal endowment of a blastocyst from the DNA of the embryonic culture medium.

The chromosomal status of the embryo from an embryo biopsy of trophoectoderm will be established (usual clinical practice), the chromosomal endowment from the DNA of the embryonic culture medium will be determined, and the results using the NICS and the conventional invasive method (Preimplantation Genetic Testing for Aneuploidy [PGT-A]) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Treatment by oocyte donation or own oocyte nd preimplantation genetic screening of aneuploidies (PGT-A).
* Embryonic cryopreservation.
* Informed consent signature

Exclusion Criteria:

* Embryo transfer without embryo freezing
* Embryonic block.
* Bad embryo quality.

Ages: 19 Years to 49 Years | Sex: Male
Age Groups: Adult
Study Population: Couples who come to the study center to carry out a PGT-A cycle. Only couples that perform treatment using their own gametes will be selected and where the indication of PGT-A will be able to be advanced maternal age, failure of implantation, repeat abortion, male factor or structural chromosomal alterations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Presence of Mosaicism | At Day 5-6 after FIV
  Presence of mosaicism
Quality value of NICS DLRS | At Day 5-6 after FIV
  Quality value of noninvasive chromosome screening (NICS) derivative Log Ratio Spread (DLRS)

CONTACTS AND LOCATIONS:
Overall Officials: Belén Lledo, PhD, Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Spain